CLINICAL TRIAL: NCT02635139
Title: Influence of Meal Skipping on Macronutrient Oxidation and Glucose Metabolism Under Isocaloric Conditions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Hohenheim (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: MealSkipping
Record Dates: First submitted 2015-12-13; First posted 2015-12-18 (Estimated); Last update posted 2017-04-25 (Actual); Status verified 2017-04

CONDITIONS: Healthy
Keywords: meal skipping; isocaloric diet; macronutrient oxidation; glucose homeostasis; arterial stiffness
MeSH Terms: conditions — Intermittent Fasting

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Breakfast Skipping (Experimental): Effect of breakfast skipping on metabolism
  Interventions: Behavioral: Breakfast skipping
- Dinner Skipping (Experimental): Effect of dinner skipping on metabolism
  Interventions: Behavioral: Dinner skipping

INTERVENTIONS:
Behavioral: Breakfast skipping — 18h fasting period in the morning
  Arms: Breakfast Skipping
Behavioral: Dinner skipping — 18h fasting period in the evening
  Arms: Dinner Skipping

SUMMARY:
Aim of the study is to investigate the impact of meal skipping (breakfast or dinner skipping) on the regulation of glucose metabolism and macronutrient balance (protein/fat/carbohydrate intake vs. -oxidation). An isoenergetic diet with 3 conventional meals (breakfast, lunch, dinner) serves as a control.

DETAILED DESCRIPTION:
The duration of the study is 7 days including 3 days with controlled diet and 4 days (including 5 nights) in a metabolic chamber at the Institute of Nutritional Medicine at the University of Hohenheim.

The study phase in the metabolic chamber consists of (i) 1 day with 3 meals/day = baseline day, (ii) 1 day with breakfast skipping, (iii) 1 day with dinner skipping, (iv) 1 washout day where the subjects leave the chamber between 7 a.m. until 7 p.m..

Beginning on the 3rd study day macronutrient and energy intake as well as the fasting periods are kept constant. To achieve comparable conditions the washout day is setted before the baseline day.

ELIGIBILITY:
Inclusion Criteria:

* healthy
* not obese (BMI<30)

Exclusion Criteria:

* food allergy
* smoking
* alternative nutrition habits
* chronic disease
* regular medication intake
* claustrophobia

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2015-12; Primary Completion 2016-07 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Regulation of glucose metabolism (substrate oxidation and insulin sensitivity) | 1 day

SECONDARY OUTCOMES:
Actigraphy-assessed sleep quality | 1 day
cardio vascular risk (lipid profile, arterial stiffness, autonomic function) | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Anja Bosy-Westphal, Prof PhD, Principal Investigator — University of Hohenheim, Stuttgart, Germany
Locations (1):
- Institute of Nutritional Medicine, University of Hohenheim, Stuttgart, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nas A, Mirza N, Hagele F, Kahlhofer J, Keller J, Rising R, Kufer TA, Bosy-Westphal A. Impact of breakfast skipping compared with dinner skipping on regulation of energy balance and metabolic risk. Am J Clin Nutr. 2017 Jun;105(6):1351-1361. doi: 10.3945/ajcn.116.151332. Epub 2017 May 10. PMID 28490511